CLINICAL TRIAL: NCT02262975
Title: A Multi-national Study to Identify Treatment Discontinuation Rate in de Novo Alzheimer's Disease Patients Who Have Been Newly Prescribed With Donepezil (Aricept) in Asia (ADOS)
Acronym: ADOS
Status: Completed | Type: Observational
Sponsor: Eisai Korea Inc. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: ART-M082-602
Record Dates: First submitted 2014-08-26; First posted 2014-10-13 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-12

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- donepezil (Aricept)

SUMMARY:
This study is an observational study conducted prospectively under routine clinical setting for 1 year with about 700 patients diagnosed as Alzheimer's disease who will be treated by donepezil (Aricept) as monotherapy. The subjects will be recruited in the selected institutions of about 8 countries in Asia.

DETAILED DESCRIPTION:
Participation in this study places no additional visit schedule, which will be determined by the investigator's judgment based on the disease progression of each subject. Investigators educate subjects to keep decided visit schedule, and collect the required information for case record from (CRF) on the visit.

ELIGIBILITY:
Inclusion Criteria:

1. Greater than or equal to 50 years old and less than 90 years old
2. Diagnosed as probable AD based on NINCDS-ADRDA
3. Patients who have been recently prescribed with donepezil (Aricept) as monotherapy
4. Patients and caregivers who signed the written informed consent from for use of personal and medical information
5. Patients with caregivers who can visit the institution together

Exclusion Criteria:

1) Patients who have taken Memantine or Acetylcholinesterase (AChE) inhibitor prior to participating in the study

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Alzheimer's disease patients who have been recently prescribed with donepezil (Aricept) as monotherapy for the first time
Sampling Method: Non-Probability Sample
Enrollment: 532 (Actual)
Dates: Start 2014-07; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Treatment discontinuation Rate | Up to 1 year

SECONDARY OUTCOMES:
Factors leading to donepezil treatment discontinuation | Up to 1 year
  Reason for the subjects who discontinued the administration of donepezil (Aricept)
Mean change in treatment duration | Up to 1 year
Percent change in treatment regimen | Up to 1 year
Mean change in the scores of cognitive assessments test | Baseline, Visit 4 [Month 6], and Visit 5: [Year 1]
Compliance of donepezil: Clinical Rating Scale (CRS) | Baseline, Visit 2 [Month 1], Visit 3 [Month 3], Visit 4 [Month 6], and Visit 5: [Year 1]
  CRS is a compliance scale ranged from 1 to 7. The higher score implies the higher compliance. 5 points or higher is defined as compliance, while 4 points or lower as non-compliance.
Compliance of donepezil: Visual Analog Scale (VAS) | Baseline, Visit 2 [Month 1], Visit 3 [Month 3], Visit 4 [Month 6], and Visit 5: [Year 1]
  VAS is a tool to determine the compliance through interview between investigators and subjects based on drug administration during previous 4 weeks. The range is from 0 to 100.

CONTACTS AND LOCATIONS:
Locations (26):
- China (6):
  - Beijing
  - Gangwon
  - Hong Kong
  - Nanjing
  - Shaanxi
  - Shanghai
- Manila, Philippines
- Singapore, Singapore
- South Korea (9):
  - Busan
  - Daegu
  - Daejeon
  - Gyeonggi-do
  - Incheon
  - Jeonju
  - Kangwon
  - Seongnam
  - Seoul
- Taiwan (7):
  - Bangkok
  - Changhua
  - Kaohsiung City
  - New Taipei City
  - Taichung
  - Tainan
  - Taipei
- Thailand (2):
  - Bangkok
  - Shanghai

REFERENCES:
- [Derived] Shim YS, Park KH, Chen C, Dominguez JC, Kang K, Kim HJ, Hong Z, Lin YT, Chu LW, Jung S, Kim S. Caregiving, care burden and awareness of caregivers and patients with dementia in Asian locations: a secondary analysis. BMC Geriatr. 2021 Apr 7;21(1):230. doi: 10.1186/s12877-021-02178-x. PMID 33827446